CLINICAL TRIAL: NCT03898024
Title: Effects of SHR-1222 on Vascular Inflammatory Factors in Patients With Low Bone Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Director, Department of Endocrinology, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019 SHR-1222
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Osteoporosis, Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): A single subcutaneous injection of SHR-1222 dose 1 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 2 (Experimental): A single subcutaneous injection of SHR-1222 dose 2 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 3 (Experimental): A single subcutaneous injection of SHR-1222 dose 3 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 4 (Experimental): A single subcutaneous injection of SHR-1222 dose 4 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo
- Cohort 5 (Experimental): A single subcutaneous injection of SHR-1222 dose 5 versus placebo
  Interventions: Drug: SHR-1222; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1222 — Pharmaceutical form: water injection; Route of administration: subcutaneous
Drug: Placebo — Pharmaceutical form: water injection; Route of administration: subcutaneous

SUMMARY:
This study aims to investigate the effects of SHR-1222 on vascular inflammatory factors in patients with low bone mass.

DETAILED DESCRIPTION:
In this study, total 50 patients with low bone mass will be enrolled and divided into 5 dose groups. In the lowest dose group 6 subjects will be recruited, among whom 4 will receive SHR-1222 and the other 2 will receive placebo. In each of the other 4 groups, 11 subjects will be recruited, among whom 9 will be administered with SHR-1222 and the other 2 with placebo.

Levels of nitric oxide (NO), Endothelin-1 (ET-1), plasminogen activator inhibitor-1 (PAI-1) and hypersensitivity C-reactive protein (hs-CRP) will be detected in patients before and after the SHR-1222 injection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Male or postmenopausal female;
* Age ≥45 and ≤59 years old;
* The body mass index (BMI) ≥18.5kg/m2 and ≤28 kg/m2;
* T value of areal bone mineral density on any lumbar spine (L1-L4) or collum femoris>-2.5 and <-1;
* The comprehensive physical examination is eligible or slightly abnormal but the researchers determine no clinical implication;
* No smoking, alcohol or drugs abuse.

Exclusion Criteria:

* Any disease affecting bone metabolism;
* Past medical history of cerebral infarction or cerebral arterial thrombosis;
* Past medical history of myocardial infarction;
* Administration of the following drugs within 6m: Hormone replacement therapy, Calcitonin Parathyroid hormone (or any derivative), Supplemental Vitamin D>1,000 IU/day, Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks before the enrollment date are allowed), Anabolic steroids, Calcitriol and available analogues, thiazide diuretics;
* Administration of the following drugs within 12m: Bisphosphonates, Fluoride for osteoporosis;
* A bone fracture within the previous 6 months;
* A lumbar spine L1-L4 or femoral neck T-score ≤-2.5;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma pancreatic acyl transferase (GGT) or total bilirubin, more than 1.5 x ULN during screening;
* 3 months prior to screening involved in any drug clinical subjects;
* Subjects determined by the researchers have any food, dietary supplement or drugs that affect SHR-1222 absorption, distribution, metabolism and excretion in 4 weeks prior to screening or within 5 half-lives;
* Serious infection, trauma or major surgery in 4 weeks prior to screening;
* A surgery plan during the study;
* Blood donation and transfusion in 3 months prior to screening;
* Unstable thyroid dysfunction in 6 months prior to screening;
* Human immunodeficiency virus antibody (HIV-ab), syphilis serological examination, hepatitis b virus surface antigen (HBsAg), hepatitis c virus antibody (HCV-ab) were positive;
* Intolerant to venous blood collection;
* A clinical history of drug allergy or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or a known allergy to experimental or similar；
* Subjects with any other situation should not be involved, which determined by the researchers.

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Assessment of serum nitric oxide (NO) change after the administration of SHR-1222 | Day0 before the administration and Day 2, 4, 7, 15, 29, 43, 57 after the administration
  NO level will be detected by nitrite/nitrate assay (colorimetric).
Assessment of serum Endothelin-1 (ET-1) change after the administration of SHR-1222 | Day0 before the administration and Day 2, 4, 7, 15, 29, 43, 57 after the administration
  ET-1 level will be detected by ELISA.
Assessment of serum plasminogen activator inhibitor-1 (PAI-1) change after the administration of SHR-1222 | Day0 before the administration and Day 2, 4, 7, 15, 29, 43, 57 after the administration
  PAI-1 level will be detected by ELISA.
Assessment of serum hypersensitivity C-reactive protein (hs-CRP) change after the administration of SHR-1222 | Day0 before the administration and Day 2, 4, 7, 15, 29, 43, 57 after the administration
  hs-CRP level will be detected by immunoturbidimetry assay.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No